CLINICAL TRIAL: NCT04749446
Title: Breast Sarcomas: A Retrospective Analysis of Clinical Features and Outcomes
Brief Title: Study on Clinical Features and Outcomes of Breast Sarcoma
Acronym: Breast-Sarc
Status: Recruiting | Type: Observational
Sponsor: Italian Sarcoma Group (Network)
Responsible Party: Sponsor
Other Study IDs: ISG-Breast-Sarc
Record Dates: First submitted 2021-02-04; First posted 2021-02-11 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Breast Sarcoma
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast sarcoma: This cohort include patients affected by breast sarcoma, referred to participating Institutions between January 2000 and June 2020.
  Interventions: Other: Treatment of Breast Sarcoma according clinical practice (includes drugs, surgery or any other received treatments)

INTERVENTIONS:
Other: Treatment of Breast Sarcoma according clinical practice (includes drugs, surgery or any other received treatments) — This observational study collects all the treatments received by the patients according clinical practices or experimental trials and therefore includes drug/biological/surgical and any other applicable treatments
  Reorder Outcome Measures

SUMMARY:
This is multi-institutional retrospective study in order to identify the most relevant clinical characteristics, treatment strategies, to explore the impact on principal clinical outcomes and finally, to suggest some principles for management and treatment of breast sarcomas.

The study will collect data about patients affected by breast sarcoma referred to participating Institutions between January 2000 and June 2020

DETAILED DESCRIPTION:
In the field of soft tissue sarcomas, breast sarcomas are a truly peculiar family of rare tumors for both their clinical history and biology of disease.

Surgery (if feasible) is the main therapeutic approach for all the patients with localized disease, while a pharmacological (chemotherapeutic) and/or radiotherapeutic treatment is reserved to those with high-risk/recurrent-relapsing/metastatic disease.

Unfortunately, there is a lack of specific prospective trials in breast sarcoma to guide the clinical decision-making and breast sarcoma patients are often sent to sarcoma referral centers only after surgery Due to sarcoma-specific clinical features, it is clear that both diagnostic and clinical strategies mandate a different approach compared to epithelial tumors. This is of key importance to reach the correct diagnosis, design the best therapeutic decision-making and subsequent follow-up.

Even if retrospective data limitations and biases, in the lack of prospective data collection, these data may be a unique and precious source of information For this reasons this multi-institutional retrospective study is aimed to identify the most relevant clinical characteristics, treatment strategies, to explore the impact on principal clinical outcomes and finally, to suggest some principles for management and treatment of breast sarcomas.

ELIGIBILITY:
Inclusion Criteria:

* >18 years at diagnosis
* primary or secondary breast sarcoma
* availability of medical data needed for the study (histopathological data, surgery, chemotherapy, including preceding chemotherapeutic regimens for secondary breast sarcomas, radiation therapy)

Exclusion Criteria:

* sarcoma metastases to the breast
* chest wall sarcomas not arising in the mammary gland
* cutaneous sarcomas

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by breast sarcma referred to participating Institutions between January 2000 and June 2020.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-04-02 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Treatments received for breast sarcoma | At diagnosis (baseline) and after 6, 12, 18, 24, 36, 48 and 60 weeks
  To describe treatment that patient diagnosed with breast sarcoma, received
Number of patients with primary breast sarcoma | Through study inclusion period, an average of 20 years
  Number of patient with a diagnosis of primary breast sarcoma

SECONDARY OUTCOMES:
Number of patients with primary breast sarcoma symptoms | Through study inclusion period, an average of 20 years
  Number of patients with primary breast sarcoma symptoms
Local-regional Relapse Free Survival (LRFS) | Every 3 months (Month 3, Month 6, Month 9...) up to 5 years
  Time elapsed form the treatment (any) start and the onset of Local-regional relapse
Progression Free Survival (PFS) | Every 3 months (Month 3, Month 6, Month 9...) up to 5 years
  Time elapsed form the treatment (any) start and the onset of progression
Overall Survival (OS) | at 5 years
  Time elapsed for the diagnosis to the death for any cause
Median time of secondary breast sarcoma presentation | Up to 3 years
  To define the median time to secondary sarcoma presentation
Impact of upfront multidisciplinary tumor board consultation | Up to 3 years
  To describe the impact of upfront multidisciplinary tumor board consultation on outcomes

CONTACTS AND LOCATIONS:
Locations (14):
- Italy (14):
  - Azienda Ospedaliera S. Orsola-Malpighi, Bologna, BO
  - Istituto Europeo di Oncologia, Milan, MI
  - Istituto Clinico Humanitas, Rozzano, MI
  - Azienda Ospedaliera Universitaria Paolo Giaccone, Palermo, PA
  - Centro di Riferimento Oncologico - Unit of Medical Oncology, Aviano, Pordenone
  - Ospedale Misericordia e Dolce, Prato, PO
  - Policlinico Universitario Campus Biomedico, Roma, RM
  - Fondazione del Piemonte per l'Oncologia IRCC Candiolo, Candiolo, Torino
  - Ospedale Umberto I, Turin, TO
  - A.O Ospedali Riuniti Marche Nord, Ancona
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Fondazione IRCCS INT Milano, Milan
  - Istituto Nazionale Tumori Regina Elena - Unit of Medical Oncology I, Roma
  - ASL Città di Torino (Dipartimento di Oncologia), Torino

IPD SHARING:
Plan to Share IPD: No
Not planned

REFERENCES:
- [Background] Al-Benna S, Poggemann K, Steinau HU, Steinstraesser L. Diagnosis and management of primary breast sarcoma. Breast Cancer Res Treat. 2010 Aug;122(3):619-26. doi: 10.1007/s10549-010-0915-y. Epub 2010 May 18. PMID 20480227
- [Background] Kirova YM, Gambotti L, De Rycke Y, Vilcoq JR, Asselain B, Fourquet A. Risk of second malignancies after adjuvant radiotherapy for breast cancer: a large-scale, single-institution review. Int J Radiat Oncol Biol Phys. 2007 Jun 1;68(2):359-63. doi: 10.1016/j.ijrobp.2006.12.011. Epub 2007 Mar 26. PMID 17379448
- [Background] Yap J, Chuba PJ, Thomas R, Aref A, Lucas D, Severson RK, Hamre M. Sarcoma as a second malignancy after treatment for breast cancer. Int J Radiat Oncol Biol Phys. 2002 Apr 1;52(5):1231-7. doi: 10.1016/s0360-3016(01)02799-7. PMID 11955733
- [Background] Sheth GR, Cranmer LD, Smith BD, Grasso-Lebeau L, Lang JE. Radiation-induced sarcoma of the breast: a systematic review. Oncologist. 2012;17(3):405-18. doi: 10.1634/theoncologist.2011-0282. Epub 2012 Feb 14. PMID 22334455
- [Background] Huang J, Mackillop WJ. Increased risk of soft tissue sarcoma after radiotherapy in women with breast carcinoma. Cancer. 2001 Jul 1;92(1):172-80. doi: 10.1002/1097-0142(20010701)92:13.0.co;2-k. PMID 11443624
- [Background] Trent II JC 2nd, Benjamin RS, Valero V. Primary soft tissue sarcoma of the breast. Curr Treat Options Oncol. 2001 Apr;2(2):169-76. doi: 10.1007/s11864-001-0059-8. PMID 12057135
- [Background] Fields RC, Aft RL, Gillanders WE, Eberlein TJ, Margenthaler JA. Treatment and outcomes of patients with primary breast sarcoma. Am J Surg. 2008 Oct;196(4):559-61. doi: 10.1016/j.amjsurg.2008.06.010. Epub 2008 Aug 23. PMID 18723152